CLINICAL TRIAL: NCT01571817
Title: Treatment of Type I Diabetes by Pancreatic Islet Transplantation Into The Gastric Submucosa
Brief Title: Pancreatic Islet Transplantation Into the Gastric Submucosa
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Andrew Posselt (Other)
Responsible Party: Sponsor-Investigator, Andrew Posselt, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Islet-Tx-Sub-DERC
Record Dates: First submitted 2012-04-03; First posted 2012-04-05 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-08

CONDITIONS: Type 1 Diabetes
Keywords: Insulin Dependent
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study intervention (Experimental): endoscopically-guided intestinal submucosal transplantation of Isolated Human Pancreatic Islets in a type 1 diabetic patient
  Interventions: Biological: Isolated Human Pancreatic Islets

INTERVENTIONS:
Biological: Isolated Human Pancreatic Islets

SUMMARY:
The overall objective of this pilot project is to evaluate the safety and efficacy of the gastric submucosal space as a novel site for clinical islet transplantation. The site has several physiologic attributes that may improve the outcomes of islet transplantation compared with the conventional intraportal transplant site.

DETAILED DESCRIPTION:
The overall objective of this pilot project is to evaluate the safety and efficacy of the gastric submucosal space as a novel site for clinical islet transplantation. Safety will be evaluated by the monitoring of side effects such as post procedural GI complications, frequency of hypo and hyperglycemic events, and immunosuppression side effects. Efficacy will be determined by accepted measures including insulin independence, long term glucose control, and reduction/elimination of hypoglycemic events.

The site has several physiologic attributes that may improve the outcomes of islet transplantation compared with the conventional intraportal transplant site.

ELIGIBILITY:
Inclusion Criteria:

Key Inclusion Criteria:

1. Primary islet allotransplant
2. Type I diabetes mellitus for a minimum of 5 years
3. One or more of the following signs or symptoms despite intensive efforts made in close cooperation with their diabetic care team:

   * Metabolic lability/instability characterized by hypoglycemia or ketoacidosis (>2 hospital admissions in the previous year), erratic glucose profiles (MAGE>120 mg/dL), or disruption in lifestyle of danger to life, self or others
   * Reduced awareness of hypoglycemia or >1 episode in the last 1.5 years of severe hypoglycemia
   * Persistently poor glucose control (as defined by HgbA1c>10% at the end of six months of Intensive management efforts with the diabetes care team)
   * Progressive secondary complications as defined by (i) a new proliferative retinopathy or clinically significant macular edema or therapy with photocoagulation during the last year; or (ii) symptomatic autonomic neuropathy (as defined by postural hypotension or neuropathic bladder)
4. Age 18 and older
5. Patients who have a renal transplant must have received their transplant at least 3 months previously and must have stable renal function (see exclusion criteria below)
6. Must be able to give written informed consent

Exclusion Criteria:

Key Exclusion Criteria:

1. Lymphopenia (<1000/µL) or leukopenia ( <3000 total leukocytes/µL)
2. Presence of panel-reactive anti-HLA antibody >20%
3. Positive lymphocytotoxic cross-match using donor lymphocytes and serum
4. Evidence of acute EBV infection (IgM>IgG) OR no serologic evidence of previous exposure to EBV (IgG>IgM)
5. Calculated or measured GFR < 50 ml/min/m2 in patients without a renal transplant.
6. Calculated or measured GFR < 40 ml/min/m2 in patients with a renal transplant.
7. Portal hypertension or history of significant liver disease
8. History of malignancy within 10 years (except for treated basal or squamous cell CA of the skin)
9. Active peptic ulcer disease or other gastric mucosal abnormalities as identified on screening endoscopy
10. Severe unremitting diarrhea or other GI disorders potentially interfering with the ability to absorb oral medications
11. Untreated proliferative retinopathy
12. Pregnancy or breastfeeding
13. Female subjects not post-menopausal or surgically sterile who are sexually active but not using an acceptable method of contraception
14. Active infections
15. Serologic evidence of infection with HIV, or HbsAg or HCV Ab positive
16. Major ongoing psychiatric illness
17. Ongoing substance abuse, drug or alcohol; or recent history of noncompliance
18. Any condition that in the opinion of the Principal Investigator does not allow safe participation in the study

    -

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Six months
  Hypo- and Hyper-glycemia limits for blood glucose related risks; during procedure, abdominal pain, duodenal hemorrhage, and duodenal perforation post-procedure, fever, cytokine release syndrome (to the thymoglobulin), immunosuppression related issues

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Posselt, M.D., Ph.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States